CLINICAL TRIAL: NCT03823430
Title: Pupillometry : Predictive Indicator in External Ventricular Drain Clamping ?
Acronym: CLAMP
Status: Completed | Type: Observational
Sponsor: Association Pro-arte (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2018-CLAMP
Record Dates: First submitted 2019-01-04; First posted 2019-01-30 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Brain Damage; External Ventricular Drain; Hydrocephalus
MeSH Terms: conditions — Brain Injuries; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pupillometry — Pupillar diameter variation measurement

SUMMARY:
Pupillar diameter variation to predict success or failure of external ventricular derivation clamping.

Pupillometry utilisation as a diagnostic tool in external ventricular clamping test in neurological ICU should improve patients care in several ways :

* earlier use of ventriculo-peritoneal or ventriculo-atrial shunts to shorten the external ventricular treatment duration and thus reduce risks of infection and hospital stay duration
* limit the medical imagery prescription and radiation exposition
* avoid neurological deterioration linked to the external ventricular drain clamping in case of the pupillometric parameters variation would be earlier than clinical signs

ELIGIBILITY:
Inclusion Criteria:

* Neurologic ICU hospitalization
* Traumatic brain injury
* External ventricular drain

Exclusion Criteria:

* Legal protection
* refusal
* therapeutics limitation
* craniectomy
* pupillar anomaly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with an external ventricular drain in neurologic ICU can be recruited in the study if all the eligibility criteria are met.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Pupillar diameter variation to predict success or failure of external ventricular clamping | 24 hours after clamping
  Pupillar diameter variation twenty-four hours after external ventricular drain clamping

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Chu Grenoble Alpes, Grenoble

IPD SHARING:
Plan to Share IPD: No